CLINICAL TRIAL: NCT00026065
Title: Hypertension: Prediction of Biofeedback Success
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01AT000310-02 (NIH); NCT00030017 (obsolete NCT alias)
Record Dates: First submitted 2001-11-09; First posted 2001-11-12 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2006-08

CONDITIONS: Essential Hypertension
Keywords: Hypertension; BIofeedback; Non-pharmacological treatment; Prediction
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Biofeedback, Psychology

INTERVENTIONS:
Behavioral: Biofeedback

SUMMARY:
Hypertension, present in more than 50 million Americans, increases the risk of cardiovascular disease and its associated complications. More persons are turning to alternative medicine to deal with their health problems. Biofeedback may reduce blood pressure and/or allow the reduction of antihypertensive medications in some patients, while having no adverse effects. Yet biofeedback therapy is time-intensive and technician-intensive. Therefore, it is critical to be able to predict which patients with essential hypertension are most likely to lower his/her blood pressure using these techniques. This research proposes to test three different means of predicting whether a hypertensive subject will or will not be successful in lowering his/her blood pressure using biofeedback. Sixty hypertensive subjects will be studied over a three-year period. The results of this study will enable those caring for hypertensive persons to recommend biofeedback in an individualized way, thereby promoting adherence.

DETAILED DESCRIPTION:
In the next century, our health care system will attempt to manage chronic illness in the largest aging population ever known. Non-adherence to pharmacological therapy and to non-pharmacological therapy will prove very costly. Hypertension, present in more than 50 million Americans, increases the risk of cardiovascular disease and its associated morbidity and mortality. Thus is it critical that adherence to treatment of hypertension be increased. While medications are effective in certain patients, their adverse effects make compliance with treatment difficult to ensure. In addition, more and more persons are turning to alternative medicine to deal with their health problems. Biofeedback offers an alternative to medical treatment, having been shown to reduce both systolic and diastolic blood pressures and/or allow the reduction of antihypertensive medications in some patients, while having no adverse effects. Yet biofeedback therapy is time-intensive and technician-intensive. Therefore, it is critical to be able to predict which patients with essential hypertension are most likely to lower his/her blood pressure using these techniques.

This research proposes to test three different means of predicting whether a hypertensive subject will or will not be successful in lowering his/her blood pressure using biofeedback. Specifically, the first set of predictive criteria to be tested is that proposed by Weaver & McGrady (1995). This model is derived from five variables: heart rate, finger temperature, forehead muscle tension, plasma rennin response to furosemide, and mean arterial pressure response to furosemide. The second prediction model is based on the magnitude of circadian variations in blood pressure as measured by 24-hour ambulatory blood pressure monitoring. The third prediction model is based on locus of control of behavior. A total of 60 hypertensive subjects will be studied over a three-year period. The results of this study will enable those caring for hypertensive persons to recommend treatment (i.e., biofeedback) in an individualized way, thereby promoting adherence.

ELIGIBILITY:
* essential hypertension
* stages 1 or 2
* not taking beta blockers or central acting alpha agonists
* permission from primary care provider

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2000-02; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn B Yucha, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Nursing, Gainesville, Florida, United States

REFERENCES:
- [Background] Yucha CB. Ambulatory blood pressure monitoring: measurement implications for research. J Nurs Meas. 2001 Spring-Summer;9(1):49-59. PMID 11469141
- [Background] Yucha CB, Clark L, Smith M, Uris P, LaFleur B, Duval S. The effect of biofeedback in hypertension. Appl Nurs Res. 2001 Feb;14(1):29-35. doi: 10.1053/apnr.2001.21078. PMID 11172227
- [Background] Weaver MT, McGrady A. A provisional model to predict blood pressure response to biofeedback-assisted relaxation. Biofeedback Self Regul. 1995 Sep;20(3):229-40. doi: 10.1007/BF01474515. PMID 7495917
- See also: Association for Applied Psychophysiology and Biofeedback — http://www.aapb.org/